CLINICAL TRIAL: NCT00588705
Title: The Communication of Genetic Risk to Adolescent Daughters of Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: 07-063
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer; Counseling
Keywords: Daughters; Communication; genetic risk; Genetic Counseling
MeSH Terms: conditions — Breast Neoplasms; Communication | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

GROUPS / COHORTS (1):
- focus group & questionaire: The group will discuss its views about how and when to talk about the risk of getting breast cancer. The focus group will be video recorded and the video recorded material will be later transcribed and carefully analyzed. In addition you will be asked to answer questions about yourself, such as education and marital status.
  Interventions: Behavioral: focus group & questionaire

INTERVENTIONS:
Behavioral: focus group & questionaire — The focus group will last about 90 minutes. However, your involvement in this study will last from the time you join until you read over the summary of what happened during the focus group and return your comments. This should be approximately 2 months. Patient will complete a questionnaire and we estimate total time for completion to be approximately 7 minutes.

SUMMARY:
The purpose of this study is to first understand how MSKCC Clinical Genetics Service doctors talk to women with breast cancer about any genetic risks they might carry, and if they help women to think about what they might say, in turn, to their relatives, especially their daughters.

A second part of the study asks women for their opinions about when and how their daughters should be told about any genetic risks.

All of this will help us develop teaching methods to help our doctors improve the way they talk about genetic risk when women with breast cancer have adolescent daughters.

ELIGIBILITY:
Inclusion Criteria:

* Women seen in the MSK CGS Service who have a diagnosis of breast cancer or
* a family history of breast cancer and
* have biological daughter(s) in the age range 12-20 years will be eligible to participate in Phase I & II.
* Women who were consented to Phase I will automatically be eligible for Phase II.

Exclusion Criteria:

* Women seen in the MSK CGS Service will be ineligible if they have no diagnosis of breast cancer and no family history of breast cancer,
* do not have a biological daughter,
* or have a biological daughter fewer than 12 or greater than 20 years(unless they were consented to Phase 1).
* Women will be ineligible if they are not English speaking,
* have intellectual or cognitive impairment,
* or active mental illness rendering them incapable of giving informed consent, such as might occur with active psychosis.

Ages: 12 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Memorial Sloan-Kettering Cancer Center (MSK) breast cancer patients seen by the clinical genetics service (CGS)and their daughters
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2007-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Is a demonstration of the effectiveness of the module in changing the behavior of clinicians after taking part in the communication skills module. | conclusion of study

SECONDARY OUTCOMES:
To examine the views of women about the provision of genetic risk information to their daughters. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Smita Banerjee, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org